CLINICAL TRIAL: NCT05158647
Title: Efficacy of Adding Magnesium Sulfate to Bupivacaine for Ilioinguinal and Iliohypogastric Nerve Block in Acute Postherniorrhaphy Pain
Brief Title: Adding Magnesium Sulfate to Bupivacaine for Ilioinguinal and Iliohypogastric Nerve Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abdelrady S Ibrahim, MD (Other)
Responsible Party: Sponsor-Investigator, Abdelrady S Ibrahim, MD, Professor Of Anesthesia and ICU, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB0000871250
Record Dates: First submitted 2021-12-03; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Magnesium Sulfate Causing Adverse Effects in Therapeutic Use
MeSH Terms: interventions — Saline Solution; Control Groups; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): 10-ml 0.5% isobaric bupivacaine and 1ml normal saline were prepared for IIIH blockade
  Interventions: Other: normal saline
- MgSo4 group (Active Comparator): 10 ml 0.5% isobaric bupivacaine and 1ml of MgSo4 10% (100 mg) were used.
  Interventions: Drug: MgSo4

INTERVENTIONS:
Other: normal saline — 10-ml 0.5% isobaric bupivacaine and 1ml normal saline were prepared for IIIH blockade
  Other Names: Control group
  Arms: control group
Drug: MgSo4 — 10 ml 0.5% isobaric bupivacaine and 1ml of MgSo4 10% (100 mg) were used
  Other Names: Magnesium Sulphate
  Arms: MgSo4 group

SUMMARY:
Regional block of ilioinguinal and iliohypogastric (IIIH) nerves has been applied to provide postoperative analgesia after inguinal hernia repair. Magnesium sulfate (MgSo4) blocks N-methyl-d-aspartate receptors, and that is why, it was used as an adjuvant to the local anesthetic (LA) in different anesthetic approaches. Although the prolongation in postoperative duration resulting from the addition of MgSO4 to LA was significant in some literature studies, it was insignificant in others. This study was designed to investigate the adjunctive effect of MgSo4 when added to bupivacaine for IIIH blockade on the postoperative analgesic duration as a primary outcome and on the verbal rating scale (VRS) scores, analgesic consumption, and hemodynamics as secondary outcomes.

DETAILED DESCRIPTION:
Regional block of ilioinguinal and iliohypogastric (IIIH) nerves has been applied to provide postoperative analgesia after inguinal hernia repair. Magnesium sulfate (MgSo4) blocks N-methyl-d-aspartate receptors, and that is why, it was used as an adjuvant to the local anesthetic (LA) in different anesthetic approaches. Although the prolongation in postoperative duration resulting from the addition of MgSO4 to LA was significant in some literature studies, it was insignificant in others. This study was designed to investigate the adjunctive effect of MgSo4 when added to bupivacaine for IIIH blockade on the postoperative analgesic duration as a primary outcome and on the verbal rating scale (VRS) scores, analgesic consumption, and hemodynamics as secondary outcomes. Patients were divided into two groups of 45 patients each by means of coded envelopes according to the LA used for IIIH blockade. In the first group (control group), patients received 10 ml 0.5% isobaric bupivacaine plus 1 ml normal saline for IIIH blockade, whereas in the second group (MgSo4 group), 10 ml 0.5% isobaric bupivacaine and 1 ml of MgSo4 10% were prepared. All the patients received intrathecal 3 ml 0.5% hyperbaric bupivacaine, and then, IIIH blockade was performed under ultrasound guidance according to the group. Postoperatively, VRS scores,analgesic duration, and any complication were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult male
* American Society of Anesthesiologists physical status I or II

Exclusion Criteria:

* Patients with body mass index greater than or equal to 35 kg/m2
* allergy to the study drugs
* on chronic analgesics or drug containing magnesium

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — adult male patients with American Society of Anesthesiologists physical status I or II, admitted to the surgical department scheduled for elective nonrelapsing unilateral inguinal herniorrhaphy under spinal anesthesia
Enrollment: 90 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Postoperative incisional pain | 2 hours postoperatively
  Postoperative incisional pain was evaluated by VRS
Postoperative incisional pain | 4 hours postoperatively
  Postoperative incisional pain was evaluated by VRS
Postoperative incisional pain | 6 hours postoperatively
  Postoperative incisional pain was evaluated by VRS
Postoperative incisional pain | 12 hours postoperatively
  Postoperative incisional pain was evaluated by VRS
Postoperative incisional pain | 18 hours postoperatively
  Postoperative incisional pain was evaluated by VRS
Postoperative incisional pain | 24 hours postoperatively
  Postoperative incisional pain was evaluated by VRS

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Elmansy, Principal Investigator — Faculty of Medicine Mansoura University
Locations (1):
- Mahmoud S Elmansy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carre P, Mollet J, Le Poultel S, Costey G, Ecoffey C. [Ilio-inguinal Ilio-hypogastic nerve block with a single puncture: an alterantive for anesthesia in emergency inguinal surgery]. Ann Fr Anesth Reanim. 2001 Aug;20(7):643-6. doi: 10.1016/s0750-7658(01)00425-7. French. PMID 11530753